CLINICAL TRIAL: NCT01414244
Title: Randomized, Placebo-Controlled Trial of Glutamine for the Treatment of Patients With Irritable Bowel Syndrome
Brief Title: Glutamine for the Treatment of Patients With Irritable Bowel Syndrome
Acronym: AT005291
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Principal Investigator, Nicholas Verne, Principal Investigator, Tulane University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-271
Record Dates: First submitted 2011-07-29; First posted 2011-08-11 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Diarrhea-Predominant Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Glutamine; Intestinal Permeability
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glutamine supplementation (Active Comparator): Glutamine
  Interventions: Drug: Glutamine
- Placebo (Placebo Comparator): Whey protein powder
  Interventions: Drug: Glutamine

INTERVENTIONS:
Drug: Glutamine — Drug
  Other Names: L-Glutamine

SUMMARY:
New and effective treatments are needed for patients with post-infectious irritable bowel syndrome (PI-IBS). We conducted a randomized, placebo-controlled trial to assess the efficacy and safety of glutamine, an abundant amino acid in the body and the principal fuel for enterocytes, in patients who developed diarrhea-predominant irritable bowel syndrome with increased intestinal permeability following an enteric infection.

DETAILED DESCRIPTION:
In a double-blind trial, eligible adults with post-infectious IBS with increased intestinal permeability were randomly assigned to receive either glutamine (5 g three times daily) or placebo for eight weeks. The primary end point was the proportion of patients who had a reduction of ≥50 on the Irritable Bowel Severity Scoring System (IBS-SS).

ELIGIBILITY:
Inclusion Criteria:

* men and women age 18-72 years old who developed post-infectious diarrhea-predominant IBS (D-IBS)
* increased intestinal permeability on Lactulose/Mannitol permeability test
* able and willing to cooperate with the study
* *absence of alcohol or NSAIDs ingestion for 2 weeks prior to inclusion into study and throughout the study duration

Exclusion Criteria:

* current participation in another research protocol or unable to give informed consent
* women with a positive urine pregnancy test or breastfeeding
* history of inflammatory bowel disease, lactose intolerance, and/or celiac sprue
* + hydrogen breath test for bacterial overgrowth
* + antiendomysial antibody titer
* use of nonsteroidal antinflammatory drug(NSAIDs) 2 weeks before or during the study
* known allergy to glutamine
* abdominal surgery except for removal of gallbladder, uterus, or appendix
* Abnormal blood urea nitrogen(BUN) and/or creatinine

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2010-11; Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: QiQi Zhou, Principal Investigator — Tulane University School of Medicine
Locations (1):
- Tulane University School of Medicine, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
Some data will be available through publications, however further plans to make all IPD available is unknown.

REFERENCES:
- [Derived] Zhou Q, Verne ML, Fields JZ, Lefante JJ, Basra S, Salameh H, Verne GN. Randomised placebo-controlled trial of dietary glutamine supplements for postinfectious irritable bowel syndrome. Gut. 2019 Jun;68(6):996-1002. doi: 10.1136/gutjnl-2017-315136. Epub 2018 Aug 14. PMID 30108163

RESULTS

PARTICIPANT FLOW:
Groups:
- Glutamine: Oral Glutamine Powder
- Placebo: Oral Whey Protein Powder
Period: Overall Study
Arm/Group | Glutamine | Placebo
Started | 54 | 52
Completed | 54 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glutamine | Placebo | Total
Number analyzed (Participants) | 54 | 52 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (9.5) | 30.9 (7.1) | 31.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 74
  Male | 17 | 15 | 32
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 54 | 52 | 106

OUTCOME MEASURES:

1. Primary Outcome: Change in the Irritable Bowel Symptom Severity Scale
Description: The primary outcome measure will be a change in the Irritable Bowel Symptom Severity Scale (IBS-SS) from baseline to 8 weeks at the conclusion of therapy. The IBS-SS scale ranges from 0 to 500 (worst). A decrease in 50 or greater in the IBS-SS is considered a positive response.
Time Frame: baseline and 8 weeks following therapy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Glutamine | Placebo
Number analyzed (Participants) | 54 | 52
units on a scale | 181 (48) | 301 (57)

2. Secondary Outcome: Intestinal Permeability
Description: The secondary outcome measure will be a change in intestinal permeability from baseline to 8 weeks at the conclusion of therapy. Intestinal permeability is measured by the urinary lactulose/mannitol ratio following ingestion of a solution of lactulose and mannitol.
Time Frame: baseline and 8 weeks following therapy
Measure: Mean (Standard Deviation); unit: lactulose/mannitol (L/M)
Arm/Group | Glutamine | Placebo
Number analyzed (Participants) | 54 | 52
lactulose/mannitol (L/M) | 0.05 (0.01) | 0.10 (0.03)

3. Secondary Outcome: Stool Frequency
Description: Baseline and 8 week at the conclusion of therapy
Time Frame: Baseline and 8 weeks following therapy
Measure: Mean (Standard Deviation); unit: stools per day
Arm/Group | Glutamine | Placebo
Number analyzed (Participants) | 54 | 52
stools per day | 2.9 (0.9) | 5.3 (2.1)

4. Secondary Outcome: Stool Consistency
Description: Bristol Stool Scale The Bristol Stool Scale characterizes stool characteristics and ranges from a minimum score of 1 with depicts hard or constipated stool to a maximum score of 7 which is watery or diarrheal stools. In this trial, stool that is less than 7 is better and depicts a good outcome.
Time Frame: Baseline and 8 weeks following therapy
Measure: Mean (Standard Deviation); unit: units on a scale (1-7)
Arm/Group | Glutamine | Placebo
Number analyzed (Participants) | 54 | 52
units on a scale (1-7) | 3.9 (1.2) | 6.6 (0.53)

ADVERSE EVENTS:
Arm/Group | Glutamine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/52
Other Adverse Events (participants affected / at risk) | 0/54 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No